CLINICAL TRIAL: NCT00995800
Title: A Double-blind, Randomised, Incomplete Block, Crossover, Placebo-controlled, Dose-response Study to Assess Bronchial Hyperresponsiveness and Airway Inflammation Effects of FlutiForm® pMDI Low and High Dose in Adult Subjects With Mild to Moderate Asthma
Brief Title: Study to Assess Airway Inflammation Effects of FlutiForm® pMDI Low and High Dose in Adults With Mild to Moderate Asthma
Acronym: FLT2503
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLT2503; 2009-009873-87
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fluticasone propionate / Formoterol fumarate (Active Comparator)
  Interventions: Drug: Fluticasone propionate / Formoterol fumarate
- Fluticasone propionate / Formoterol fumarate placebo (Placebo Comparator)
  Interventions: Drug: Fluticasone propionate / Formoterol fumarate

INTERVENTIONS:
Drug: Fluticasone propionate / Formoterol fumarate — 2 dose strength vs. placebo

SUMMARY:
This is a dose-response study to determine how various measurements of airway inflammation respond to high and low dose FlutiForm®, and compared to placebo.

DETAILED DESCRIPTION:
The study consists of two 4-week treatment periods, each preceded by a 14-21 wash-out period. Subjects will be randomised to receive two of the three study treatments - FlutiForm® pMDI 50/5 µg, FlutiForm® pMDI 250/10 µg, or placebo (dummy inhaler). During the wash-out periods, subjects will take only salbutamol, if required, as rescue medication.

Subjects will record a daily diary for PEFR, study medication use, rescue medication use, asthma symptom scores, and sleep disturbance due to asthma. Assessments performed at study clinic visits include inhaled adenosine 5'-monophosphate (AMP) challenge test, induced sputum test, exhaled nitric oxide (eNO) test, and spirometry tests. Safety will be assessed by lab tests, vital signs, ECG and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 18 and 55 years inclusive.
2. Females less than one year post-menopausal must have a negative serum or urine pregnancy test recorded at the screening visit prior to the first dose of study medication in each treatment period, be non-lactating, and be willing to use adequate and highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device, hormonal), sexual abstinence or vasectomised partner.
3. Known history of mild to moderate asthma for ≥ 6 months prior to the screening visit.
4. Subject has not received systemic (injectable or oral) corticosteroid medication in the 12 weeks prior to the study screening visit.
5. Demonstrate a FEV1 of ≥ 60% predicted FEV1 (Quanjer et al, 1993) at the screening visit, following appropriate withholding of asthma medications (no long-acting β2-agonist or short-acting β2-agonist/anticholinergic use 12 hours and 6 hours prior to screening, respectively).
6. Demonstrate AMP challenge PC20FEV1 < 60 mg/mL, following appropriate withholding of asthma medication (no short-acting bronchodilator use 6 hours prior to the AMP challenge test at Visit 2).
7. Non-smoker for at least 12 months prior to study screening. Ex-smokers must have a smoking history equivalent to less than "10 pack years" (i.e. at least 1 pack of 20 cigarettes per day for 10 years or 10 packs per day for 1 year, etc.).
8. Demonstrate satisfactory technique in the use of the pMDI.
9. Willing and able to enter information in the diary and attend all study visits.
10. Willing and able to substitute study medication for their pre-study prescribed asthma medication for the duration of the study.
11. Written informed consent obtained.

Exclusion Criteria:

1. Near fatal or life-threatening (including intubation) asthma within the past year.
2. Hospitalisation or an emergency visit for asthma within 4 weeks prior to the screening visit.
3. History of omalizumab use within the past 6 months.
4. Current evidence or history of any clinically significant disease or abnormality including uncontrolled coronary artery disease, congestive heart failure, myocardial infarction, or cardiac dysrhythmia. 'Clinically significant' is defined as any disease that, in the opinion of the Investigator, would put the subject at risk through study participation, or which would affect the outcome of the study.
5. In the investigator's opinion a clinically significant upper or lower respiratory infection within 4 weeks prior to the screening visit.
6. Significant, non-reversible, active pulmonary disease (e.g. chronic obstructive pulmonary disease (COPD), cystic fibrosis, bronchiectasis, tuberculosis).
7. Known Human Immunodeficiency Virus (HIV)-positive status.
8. Current evidence or history of alcohol and/or substance abuse within 12 months prior to the screening visit.
9. Subjects who have taken beta-blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, astemizole (Hismanal), quinidine type antiarrhythmics, or potent CYP 3A4 inhibitors such as ketoconazole within one week prior to the screening visit.
10. History of leukotriene receptor antagonist use, e.g. montelukast, within one week prior to the screening visit.
11. Current use of medications other than those allowed in the protocol that will have an effect on bronchospasm and/or pulmonary function.
12. Anti-histamines within 2 weeks prior to the screening visit; non-steroidal anti-inflammatory drugs, oral decongestants, inhaled cromolyn sodium, nedocromil sodium within one week prior to the screening visit.
13. Current evidence or history of hypersensitivity or idiosyncratic reaction to test medications, rescue medication, or components.
14. Use of an investigational drug within 30 days prior to the screening visit (12 weeks if an oral or injectable steroid).
15. Current participation in a clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Effects of each dose strength on bronchial hyperresponsiveness to inhaled adenosine 5'-monophosphate (AMP) challenge.

SECONDARY OUTCOMES:
eNO, % of eosinophils in induced sputum, comp each dose placebo of bronchial hyperresponsive to AMP challenge. Lung func, rescue med use, asthma symps,& exacerbations sleep disturbance, discon due to lack of efficacy & spontaneously reported AEs.

CONTACTS AND LOCATIONS:
Locations (1):
- KLB, Lübeck, Germany

REFERENCES:
- See also: Results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=FLT2503